CLINICAL TRIAL: NCT04591600
Title: Controlled Randomized Clinical Trial on Using Ivermectin With Doxycycline for Treating COVID-19 Patients in Baghdad, Iraq
Brief Title: Effectiveness of Ivermectin and Doxycycline on COVID-19 Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alkarkh Health Directorate-Baghdad (Other Government)
Responsible Party: Principal Investigator, Ahmed Sahib Abdulamir, M.B.Ch.,B., Phd Virology, Professor, Alkarkh Health Directorate-Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVM-DOX
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: Ivermectin; Doxycycline; COVID-19; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Ivermectin; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin-Doxycycline (Experimental): Ivermectin 200ug/kg PO per day for two days, and in some patients who needed more time to recover, a third dose 200ug/kg PO per day was given 7 days after the first dose. Doxycycline 100mg capsule PO every 12h per day was given for 5-10 days, based on the clinical improvement of patients. In addition, standard of care was given to the patients of Ivermectin-Doxycycline group based on the clinical condition of each patient.
  Interventions: Drug: Ivermectin and Doxycyline; Drug: Standard of care
- Control (Active Comparator): Control group: The patients in this group received only standard care which included all or some of the following, according to the clinical condition of each patient.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Ivermectin and Doxycyline — Ivermectin 200ug/kg PO per day for two days, and in some patients who needed more time to recover, a third dose 200ug/kg PO per day was given 7 days after the first dose. Doxycycline 100mg capsule PO every 12h per day was given for 5-10 days, based on the clinical improvement of patients. In addition, standard care was given to the patients of Ivermectin-Doxycycline group based on the clinical condition of each patient.
  Other Names: Stromectol and Doxycin
  Arms: Ivermectin-Doxycycline
Drug: Standard of care — Standard care
  * Acetaminophen 500mg on need
  * Vitamin C 1000mg twice/ day
  * Zinc 75-125 mg/day
  * Vitamin D3 5000IU/day
  * Azithromycin 250mg/day for 5 days
  * Oxygen therapy/ C-Pap if needed
  * dexamethasone 6 mg/day or methylprednisolone 40mg twice per day, if needed
  * Mechanical ventilation, if needed
  Other Names: Control arm

SUMMARY:
A randomized controlled trial on using Ivermectin and doxycycline to treat mild-moderate outpatients, severe, and critical inpatients of Coronavirus disease 19 (COVID-19) along with standard of care. Seventy Iraqi COVID-19 patients received Ivermectin and Doxycycline plus standard of care versus seventy Iraqi COVID-19 patients received standard of care only. .

DETAILED DESCRIPTION:
Objectives: COVID-19 patients suffer from the lack of curative therapy. Hence, there is an urgent need to try old re-purposed drugs on COVID-19. Methods: Randomized controlled study on 70 COVID-19 patients (48 mild-moderate, 11 severe, and 11 critical patients) treated with 200ug/kg PO of Ivermectin per day for 2 days along with 100mg PO doxycycline twice per day for 5-10 days plus standard therapy; the second arm is 70 COVID-19 patients (48 mild-moderate and 22 severe and zero critical patients) on standard therapy. The time to recovery, the progression of the disease, and the mortality rate were the outcome-assessing parameters.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients at any stage of this disease

Exclusion Criteria:

* Patients of allergic history to Ivermectin or to doxycyline

Ages: 16 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Mortality rate | Up to 8 weeks
  The effect of the experimental drugs to reduce the mortality rate (death rate) of treated patients
Rate of progression disease | up to 8 weeks
  rate of patients under treatment who undergo progression of disease to a more advanced stage

SECONDARY OUTCOMES:
Time to recovery | Up to 8 weeks
  time needed by treated patients to recover (become symptoms free and polymerase chain reaction, or PCR, negative)

CONTACTS AND LOCATIONS:
Locations (1):
- Akarkh Healt hdirectorate, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No